CLINICAL TRIAL: NCT07079722
Title: Educational Program for Type 2 Diabetes Prevention With Integrated Physical Exercise: Digital and In-Person Approach
Brief Title: More Health Less Diabetes
Acronym: MHLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHLD FMH
Record Dates: First submitted 2025-05-23; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-05

CONDITIONS: Pre-diabetes
Keywords: Diabetes; Exercise; Community programs; Prevention; Health
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The "More Health, Less Diabetes" research project is a randomized controlled trial (RCT) with three distinct groups: a control group (CG), an online intervention group (OIG), and an in-person intervention group (IIG). The OIG will receive online educational sessions and structured home-based exercises, while the IIG will participate in in-person educational sessions and supervised physical exercise. The control group will not participate in educational sessions or structured physical exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Active Comparator): The control group will not participate in educational sessions or structured physical exercise.
  Interventions: Behavioral: Exercise
- In-person intervention group (IIG). (Experimental): The IIG will participate in in-person educational sessions and supervised physical exercise
  Interventions: Behavioral: Exercise
- Online intervention group (OIG) (Experimental): The OIG will receive online educational sessions and structured home-based exercises
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — This project is a randomized controlled trial (RCT) with three distinct groups: a control group (CG), an online intervention group (OIG), and an in-person intervention group (IIG). The OIG will receive online educational sessions and structured home-based exercises, while the IIG will participate in in-person educational sessions and supervised physical exercise. The control group will not participate in educational sessions or structured physical exercise.

SUMMARY:
The "More Health, Less Diabetes" project is a hybrid randomized controlled trial to prevent type 2 diabetes in individuals at risk through structured exercise and lifestyle education. While exercise benefits for people with diabetes are well-documented, evidence remains limited on the effectiveness and cost-effectiveness of in-person and home-based exercise programs in a prediabetic population. This study aims to understand the clinical and cost-effectiveness of a three-arm RCT (online, in-person, and a control group) in people at high risk of developing T2DM. This 12-month program includes six months of supervised exercise (3 times/week) and a six-month follow-up. During the first six months, both intervention groups will attend educational sessions to improve health literacy and promote healthy habits. The primary outcome will be 2h glycemia in an oral glucose tolerance test. Secondary outcomes include other aspects of glycemic control (HbA1c, fasting glycemia, HOMA-IR, Matsuda index), 24-hour movement, body composition, vascular health, physical fitness, and cost-effectiveness using a social return on investment approach.

DETAILED DESCRIPTION:
Introduction

Diabetes is a major public health concern affecting approximately 11.1% of the adult population (588.7 million people), with projections suggesting an increase to 852 million by 2050. In Portugal, diabetes affects approximately 14.1% of the population between 20-79 years, with an additional 28.6% of the Portuguese population having intermediate hyperglycemia. These alarming values result in a financial burden for the Portuguese healthcare system, with annual costs ranging between 6-7% of total Portuguese healthcare cost.

On this note, there is evidence that 70% of people with intermediate hyperglycemia tend to develop type 2 diabetes mellitus (T2DM) in a 10- year follow-up . Risk factors, such as higher BMI and waist circumference values, physical inactivity, unhealthy diet, and poor health literacy, are directly associated with the development of T2DM. Furthermore, from the early stages of pre-diabetes, there is strong evidence of structural and functional vascular changes, which are known to increase in the medium to long/term micro and macrovascular complications.

From an economic and public health perspective, exercise interventions in a community setting are worth investing for T2DM management and prevention. The Diabetes Prevention Program (DPP) reported that 5-7% individuals who met the physical activity goals reduced their incidence of T2DM by 44% - even without weight loss. The 15-year follow-up study of the DPP has also provided evidence of the superior impact of a lifestyle intervention for preventing the development of DMT2 compared to just medication. Furthermore, our group has also shown the importance of exercise in improving health-related biomarkers in people with T2DM. Despite its known benefits, evidence suggests that comparability across exercise interventions is limited due to several issues, such as heterogeneity in intervention type, design, and delivery. For instance, studies have explored the impact of online or in-person regimes to address how lifestyle interventions should be delivered. The current body of literature on online interventions suggests that the improvements in health-related outcomes and adherence may be compromised in the medium to long term. However, online interventions are known to be more scalable and less expensive than in-person programs. On the other hand, evidence from national in-person programs, such as the "Diabetes em Movimento" program, has shown that community-based exercise programs can significantly improve cardiometabolic parameters and still be cost-effective in people with T2DM. This program is currently implemented in 52 Portuguese municipalities. Despite the effectiveness and cost-effectiveness of such exercise programs on the T2DM population, there is a gap of experimental evidence of how in-person or online lifestyle programs impact those at risk of developing T2DM. Thus, it is crucial to develop a proof-of-concept, evidence-based exercise program tailored to individuals at risk of T2DM that can ultimately be scaled to reduce the burden of T2DM at a population level. Implementing a hybrid randomized controlled trial would allow for a comprehensive cost- effectiveness evaluation, helping to determine whether online or in-person delivery yields the most economically viable and clinically beneficial outcomes.

Aims

1. To analyze the clinical effectiveness of a 6-month online regime vs. in-person lifestyle intervention vs. controls on post-prandial 2h glucose in an OGTT in people at an increased risk of developing type 2 diabetes and its impact at a 12-month follow-up period.

Secondary:

1. To evaluate the cost-effectiveness of the intervention with exercise and educational sessions, using a social return on investment approach (SROI) in an online regime vs. an in-person regime vs. a control group at the 6-month and 12-month periods
2. Assess differences at the 6-month intervention and 12-month follow-up period in other aspects of glycemic control (HOMA-IR, Matsuda index), body composition regional and total outcomes, structural and functional vascular health, handgrip strenght, 24-hour movement variables, and quality of life in the different intervention arms (e.g., In-person, online, and control).

Recruitment

Participants will be recruited for an interventional study targeting individuals with prediabetes or a high-to-very-high risk of Type 2 Diabetes, based on risk stratification using the FINDRISC questionnaire. Recruitment will take place through primary healthcare consultations in the Oeiras municipality. Individuals diagnosed with Diabetes Mellitus, those who underwent a diabetes risk assessment more than three years ago, or those with a confirmed diagnosis of diabetes will be excluded. Power calculations and sample size estimation (G-Power, Version 3.1.3) were based on an effect size of 0.2 for the Finnish Diabetes Risk Score (FINDRISC), with α = 0.05 and a power of 0.80. The final sample will consist of 90 participants, accounting for an expected dropout rate of 30%.

Study Design

The "More Health, Less Diabetes" research project is a randomized controlled trial (RCT) with three distinct groups: a control group (CG), an online intervention group (OIG), and an in-person intervention group (IIG). The OIG will receive online educational sessions and structured home-based exercises, while the IIG will participate in in-person educational sessions and supervised physical exercise. The control group will not participate in educational sessions or structured physical exercise.

The intervention will last six months across all groups, with additional follow-up assessments at 12 months. No educational sessions will occur during the follow-up period, and exercise will be optional for all groups. During this phase, control group participants may also join exercise sessions.

Randomization will be automated and conducted by a team member not directly involved in data collection or intervention processes. The Redcap® platform will be used for randomization, ensuring a 1:1:1 allocation ratio stratified by age.

Laboratory Analyses

Biochemical assessments will be conducted through primary healthcare centers. Participants will undergo clinical analyses of glycated hemoglobin (HbA1c) and fasting blood glucose, as well as a 2-hour glucose tolerance test (OGTT) after ingesting 75g of glucose at baseline, after six months, and after one year.

Anthropometric Measurements

Participants' weight and height will be measured with a precision of 0.01 kg and 0.1 cm, respectively, using a scale with an integrated stadiometer (Seca, Hamburg, Germany). Body Mass Index (BMI) will be calculated using the formula [weight (kg)/height² (m²)]. Measurements will be collected at baseline, six months, and one year.

Bioelectrical Impedance Analysis

Whole-body bioelectrical impedance analysis (BIA) will be performed using the AKERN BIA 101/BIVA PRO device, a phase-sensitive single-frequency BIA device. Participants will be instructed to lie down for 10 minutes before measurement. After cleaning the skin, eight low-impedance electrodes (Biatrodes, Akern Srl, Florence, Italy) will be placed on the dorsal surfaces of the feet, ankles, wrists, and hands. This analysis will be performed at baseline, after six months, and after one year.

Dual-Energy X-ray Absorptiometry (DXA)

Lean body mass and fat mass will be determined for the whole body and regionally using dual-energy X-ray absorptiometry (DXA; Hologic Explorer W, QDR for Windows version 12.4, Waltham, MA, USA). This evaluation will be conducted at baseline, after six months, and after one year.

Maximal Cardiopulmonary Exercise Testing

A maximal cardiopulmonary exercise test will be used to assess peak aerobic capacity, peak power output (PPO), and pre-existing cardiac conditions. A ramp incremental protocol will be performed to exhaustion on a cycle ergometer (Monark 839E, Kroons Vag, Sweden). Workload will start at 20 Watts/min and increase in increments of 5-20 Watts/min, based on individual cardiopulmonary responses in the first minute, with a constant cadence of 60 rpm. A cardiologist will monitor all tests using a 12-lead electrocardiogram, and additional data, including heart rate, will be recorded using Omnia software (Cosmed, Rome, Italy). Expired and inspired gases will be continuously analyzed using a Quark RMR w/CPET gas analyzer (version 9.1, Cosmed, Rome, Italy).

Handgrip Strength

The handgrip strength will be accessed using a dynamometer (JAMAR), which measures the upper limb strength and can estimate an individual's total strength.

Vascular Health

Vascular functional health will be measured via pulse wave velocity on the carotid-femoral, carotid-radial, and femoral dorsalis sites (Complior, Alam Medical, France). Structural indices will be assessed via intima-media thickness and arterial stiffness using ultrasonography of the right common carotid artery (Arietta V60, Hitachi Aloka, Japan).

ELIGIBILITY:
Inclusion Criteria:

1. High or Very High Risk according to the FINDRISC questionnaire;
2. Analytical confirmation of no diagnostic criteria for Diabetes, following a type 2 Diabetes risk assessment;
3. Committed to making lifestyle changes to manage diabetes;
4. Internet access;
5. Availability to participate in the program as required (schedule, location);

Exclusion Criteria:

1. pregnancy (self-report/medical record);
2. Inability to use digital devices
3. Presence of abnormalities on exercise stress test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
2-hour glucose tolerance test (OGTT) | 1 year
  Biochemical assessments will be conducted through primary healthcare centers. Participants will undergo clinical analyses of a 2-hour glucose tolerance test (OGTT) after ingesting 75g of glucose at baseline, after six months, and after one year.

SECONDARY OUTCOMES:
Height in centimeters | 1 year
  Participants' height will be measured with a precision of 0.1 cm, using a scale with an integrated stadiometer (Seca, Hamburg, Germany). Measurements will be collected at baseline, six months, and one year.
Weight in kilograms | 1 year
  Participants' weight will be measured with a precision of 0.01 kg, using a scale with an integrated stadiometer (Seca, Hamburg, Germany). Measurements will be collected at baseline, six months, and one year.
Body Mass Index | 1 year
  Body Mass Index (BMI) will be calculated using the formula [weight (kg)/height² (m²)]. Measurements will be collected at baseline, six months, and one year.
Effectiveness of the program | Through study completion, an average of 1 year
  The primary effectiveness outcome will be the change in 2-hour glucose OGTT levels.
Costs of the program | Through study completion, an average of 1 year
  The total cost of the program will be calculated by summing direct costs (e.g., facility use, instructor fees, and equipment) and indirect costs (e.g., participant time and transportation, where applicable).
Cost-effectiveness | Through study completion, an average of 1 year
  Cost-effectiveness will be assessed using the Social Return on Investment framework, which estimates the social value generated for each monetary unit invested. This outcome measure will combine cost and effectiveness of the program.
Glycated Hemoglobin | 1 year
  Biochemical assessments will be conducted through primary healthcare centers. Participants will undergo clinical analyses of glycated hemoglobin (HbA1c).Measurements will be collected at baseline, six months, and one year.
Fasting blood glucose | 1 year
  Biochemical assessments will be conducted through primary healthcare centers. Participants will undergo clinical analyses of fasting blood glucose. Measurements will be collected at baseline, six months, and one year.
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | 1 year
  HOMA-IR will be calculated to estimated insulin resistance. Measurements will be collected at baseline, six months, and one year.
Matsuda Index | 1 year
  Matsuda Index will be calculated to assess insulin sensitivity. Measurements will be collected at baseline, six months, and one year.
Bioelectrical Impedance Analysis | 1 year
  Whole-body bioelectrical impedance analysis (BIA) will be performed using the AKERN BIA 101/BIVA PRO device, a phase-sensitive single-frequency BIA device. Participants will be instructed to lie down for 10 minutes before measurement. After cleaning the skin, eight low-impedance electrodes (Biatrodes, Akern Srl, Florence, Italy) will be placed on the dorsal surfaces of the feet, ankles, wrists, and hands. This analysis will be performed at baseline, after six months, and after one year.
Maximal Cardiopulmonary Exercise Testing | 1 year
  A maximal cardiopulmonary exercise test will be used to assess peak aerobic capacity, peak power output (PPO), and pre-existing cardiac conditions. A ramp incremental protocol will be performed to exhaustion on a cycle ergometer (Monark 839E, Kroons Vag, Sweden). Workload will start at 20 Watts/min and increase in increments of 5-20 Watts/min, based on individual cardiopulmonary responses in the first minute, with a constant cadence of 60 rpm. A cardiologist will monitor all tests using a 12-lead electrocardiogram, and additional data, including heart rate, will be recorded using Omnia software (Cosmed, Rome, Italy). Expired and inspired gases will be continuously analyzed using a Quark RMR w/CPET gas analyzer (version 9.1, Cosmed, Rome, Italy). Measurements will be collected at baseline, six months, and one year.
Dual-Energy X-ray Absorptiometry (DXA) | 1 year
  Lean body mass and fat mass will be determined for the whole body and regionally using dual-energy X-ray absorptiometry (DXA; Hologic Explorer W, QDR for Windows version 12.4, Waltham, MA, USA). This evaluation will be conducted at baseline, after six months, and after one year.
Handgrip Strenght | 1 year
  The handgrip strength will be accessed using a dynamometer (JAMAR), which measures the upper limb strength and can estimate an individual's total strength. Measurements will be collected at baseline, six months, and one year.
Vascular Health-pulse wave velocity | 1 year
  Vascular functional health will be measured via pulse wave velocity on the carotid-femoral, carotid-radial, and femoral dorsalis sites (Complior, Alam Medical, France). Measurements will be collected at baseline, six months, and one year.
Vascular structural indices- Arterial Stiffness | 1 year
  Structural indices will be assessed viaarterial stiffness using ultrasonography of the right common carotid artery (Arietta V60, Hitachi Aloka, Japan). Measurements will be collected at baseline, six months, and one year.
Vascular structural indices- Intima-media thickness | 1 year
  Structural indices will be assessed via intima-media thickness using ultrasonography of the right common carotid artery (Arietta V60, Hitachi Aloka, Japan). Measurements will be collected at baseline, six months, and one year.
GRAFFAR Questionnaire | 1 year
  GRAFFAR questionnaire will be used to assess the socioeconomic status of the participants. Measurements will be collected at baseline, six months, and one year.
FINDRISC Questionnaire | 1 year
  FINDRISC questionnaire will be used to assess participants' risk of developing type 2 diabetes. Measurements will be collected at baseline, six months, and one year.
EQ-5D-5L Questionnaire | 1 year
  EQ-5D-5L questionnaire will be used to assess participants' quality of life. Measurements will be collected at baseline, six months, and one year.
IPAQ Questionnaire | 1 year
  Adapted IPAQ questionnaire will be used to assess participants' physical activity level. Measurements will be collected at baseline, six months, and one year.
PREDIMED Questionnaire | 1 year
  PREDIMED questionnaire will be used to assess participants' diet. Measurements will be collected at baseline, six months, and one year.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Human Kinetics, Lisbon, Lisbon District, Portugal

REFERENCES:
- [Background] Diabetes Prevention Program Research Group. Long-term effects of lifestyle intervention or metformin on diabetes development and microvascular complications over 15-year follow-up: the Diabetes Prevention Program Outcomes Study. Lancet Diabetes Endocrinol. 2015 Nov;3(11):866-75. doi: 10.1016/S2213-8587(15)00291-0. Epub 2015 Sep 13. PMID 26377054
- [Background] Magliano DJ, Boyko EJ; IDF Diabetes Atlas 10th edition scientific committee. IDF DIABETES ATLAS [Internet]. 10th edition. Brussels: International Diabetes Federation; 2021. Available from http://www.ncbi.nlm.nih.gov/books/NBK581934/ PMID 35914061
- [Background] Al Ozairi E, Alsaeed D, Al Roudhan D, Jalali M, Mashankar A, Taliping D, Abdulla A, Gill JMR, Sattar N, Welsh P, Gray SR. The effect of home-based resistance exercise training in people with type 2 diabetes: A randomized controlled trial. Diabetes Metab Res Rev. 2023 Oct;39(7):e3677. doi: 10.1002/dmrr.3677. Epub 2023 Jun 17. PMID 37330638
- [Background] Dunstan DW, Daly RM, Owen N, Jolley D, Vulikh E, Shaw J, Zimmet P. Home-based resistance training is not sufficient to maintain improved glycemic control following supervised training in older individuals with type 2 diabetes. Diabetes Care. 2005 Jan;28(1):3-9. doi: 10.2337/diacare.28.1.3. PMID 15616225
- [Background] Dunstan DW, Vulikh E, Owen N, Jolley D, Shaw J, Zimmet P. Community center-based resistance training for the maintenance of glycemic control in adults with type 2 diabetes. Diabetes Care. 2006 Dec;29(12):2586-91. doi: 10.2337/dc06-1310. PMID 17130189
- [Background] Golovaty I, Wadhwa S, Fisher L, Lobach I, Crowe B, Levi R, Seligman H. Reach, engagement and effectiveness of in-person and online lifestyle change programs to prevent diabetes. BMC Public Health. 2021 Jul 5;21(1):1314. doi: 10.1186/s12889-021-11378-4. PMID 34225674
- [Background] Correia IR, Hetherington-Rauth M, Magalhaes JP, Judice PB, Rosa GB, Henriques-Neto D, Manas A, Ara I, Silva AM, Sardinha LB. Compensatory mechanisms from different exercise intensities in type 2 diabetes: a secondary analysis of a 1-year randomized controlled trial. Acta Diabetol. 2023 May;60(5):645-654. doi: 10.1007/s00592-023-02038-7. Epub 2023 Feb 2. PMID 36729308
- [Background] Magalhaes JP, Hetherington-Rauth M, Judice PB, Correia IR, Rosa GB, Henriques-Neto D, Melo X, Silva AM, Sardinha LB. Interindividual Variability in Fat Mass Response to a 1-Year Randomized Controlled Trial With Different Exercise Intensities in Type 2 Diabetes: Implications on Glycemic Control and Vascular Function. Front Physiol. 2021 Sep 16;12:698971. doi: 10.3389/fphys.2021.698971. eCollection 2021. PMID 34603073
- [Background] Mendes R, Sousa N, Reis VM, Themudo-Barata JL. Implementing Low-Cost, Community-Based Exercise Programs for Middle-Aged and Older Patients with Type 2 Diabetes: What Are the Benefits for Glycemic Control and Cardiovascular Risk? Int J Environ Res Public Health. 2017 Sep 13;14(9):1057. doi: 10.3390/ijerph14091057. PMID 28902144
- [Background] Magalhaes JP, Melo X, Correia IR, Ribeiro RT, Raposo J, Dores H, Bicho M, Sardinha LB. Effects of combined training with different intensities on vascular health in patients with type 2 diabetes: a 1-year randomized controlled trial. Cardiovasc Diabetol. 2019 Mar 18;18(1):34. doi: 10.1186/s12933-019-0840-2. PMID 30885194
- [Background] Magalhaes JP, Judice PB, Ribeiro R, Andrade R, Raposo J, Dores H, Bicho M, Sardinha LB. Effectiveness of high-intensity interval training combined with resistance training versus continuous moderate-intensity training combined with resistance training in patients with type 2 diabetes: A one-year randomized controlled trial. Diabetes Obes Metab. 2019 Mar;21(3):550-559. doi: 10.1111/dom.13551. Epub 2018 Oct 29. PMID 30284352
- [Background] Hetherington-Rauth M, Magalhaes JP, Judice PB, Melo X, Sardinha LB. Vascular improvements in individuals with type 2 diabetes following a 1 year randomised controlled exercise intervention, irrespective of changes in cardiorespiratory fitness. Diabetologia. 2020 Apr;63(4):722-732. doi: 10.1007/s00125-020-05089-5. Epub 2020 Jan 20. PMID 31960071
- [Background] Magalhaes JP, Santos DA, Correia IR, Hetherington-Rauth M, Ribeiro R, Raposo JF, Matos A, Bicho MD, Sardinha LB. Impact of combined training with different exercise intensities on inflammatory and lipid markers in type 2 diabetes: a secondary analysis from a 1-year randomized controlled trial. Cardiovasc Diabetol. 2020 Oct 7;19(1):169. doi: 10.1186/s12933-020-01136-y. PMID 33028418
- [Background] Hamman RF, Wing RR, Edelstein SL, Lachin JM, Bray GA, Delahanty L, Hoskin M, Kriska AM, Mayer-Davis EJ, Pi-Sunyer X, Regensteiner J, Venditti B, Wylie-Rosett J. Effect of weight loss with lifestyle intervention on risk of diabetes. Diabetes Care. 2006 Sep;29(9):2102-7. doi: 10.2337/dc06-0560. PMID 16936160
- [Background] Barbosa A, Brito J, Figueiredo P, Seabra A, Ding D, Mendes R. How much does it cost to implement a community-based walking football programme for patients with type 2 diabetes? BMJ Open Sport Exerc Med. 2023 Jun 7;9(2):e001549. doi: 10.1136/bmjsem-2023-001549. eCollection 2023. PMID 37304893
- [Background] Green DJ, Hopman MT, Padilla J, Laughlin MH, Thijssen DH. Vascular Adaptation to Exercise in Humans: Role of Hemodynamic Stimuli. Physiol Rev. 2017 Apr;97(2):495-528. doi: 10.1152/physrev.00014.2016. PMID 28151424
- [Background] Wasserman DH, Wang TJ, Brown NJ. The Vasculature in Prediabetes. Circ Res. 2018 Apr 13;122(8):1135-1150. doi: 10.1161/CIRCRESAHA.118.311912. PMID 29650631
- [Background] Ligthart S, van Herpt TT, Leening MJ, Kavousi M, Hofman A, Stricker BH, van Hoek M, Sijbrands EJ, Franco OH, Dehghan A. Lifetime risk of developing impaired glucose metabolism and eventual progression from prediabetes to type 2 diabetes: a prospective cohort study. Lancet Diabetes Endocrinol. 2016 Jan;4(1):44-51. doi: 10.1016/S2213-8587(15)00362-9. Epub 2015 Nov 11. PMID 26575606
- [Background] Beulens J, Rutters F, Ryden L, Schnell O, Mellbin L, Hart HE, Vos RC. Risk and management of pre-diabetes. Eur J Prev Cardiol. 2019 Dec;26(2_suppl):47-54. doi: 10.1177/2047487319880041. PMID 31766914
- [Background] Diabetologia SPd. Diabetes: Factos e Números- O ano de 2019, 2020 e 2021- Relatório Anual do Observatório Nacional de Diabetes. 2023.